CLINICAL TRIAL: NCT00238225
Title: A Phase I Study of Oral Calcitriol in Combination With Ketoconazole in Refractory Advanced Malignancies
Brief Title: Calcitriol, Ketoconazole, and Dexamethasone in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Purpose: Treatment
Other Study IDs: I 33204; RPCI-I-33204
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Calcitriol; Dexamethasone; Ketoconazole

INTERVENTIONS:
Dietary Supplement: calcitriol
Drug: dexamethasone
Drug: ketoconazole

SUMMARY:
RATIONALE: Calcitriol may cause solid tumor cells to look more like normal cells, and to grow and spread more slowly. Ketoconazole and dexamethasone may help calcitriol work better by making tumor cells more sensitive to the drug. Giving calcitriol together with ketoconazole and dexamethasone may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of calcitriol when given together with ketoconazole and dexamethasone in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of calcitriol when administered with ketoconazole and dexamethasone in patients with metastatic or unresectable solid tumors.

Secondary

* Determine the tolerability and toxic effects of this regimen in these patients.
* Determine tumor response in patients treated with this regimen.
* Determine the pharmacokinetics of calcitriol and dexamethasone with or without ketoconazole in these patients.
* Determine the pharmacodynamics of this regimen, in terms of CYP24 expression and activity and vitamin D receptor expression in peripheral blood mononuclear cells, in these patients.

OUTLINE: This is a dose-escalation study of calcitriol.

Patients receive oral dexamethasone twice daily beginning on day 0 and oral ketoconazole 3 times daily beginning on day 4. Patients also receive oral calcitriol once daily on days 1-3 of each week. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of calcitriol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed for up to 30 days.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Metastatic or unresectable disease
* Standard curative or reliable palliative therapy is no longer effective OR does not exist
* Brain metastases allowed provided they have been treated with surgery or radiotherapy AND are stable

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 75,000/mm^3

Hepatic

* AST/ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* No unstable or uncompensated hepatic disease

Renal

* Creatinine ≤ 2 mg/dL
* No unstable or uncompensated renal disease
* No history of kidney, urethral, or bladder stones within the past 5 years

Cardiovascular

* Ejection fraction ≥ 30%
* No symptomatic congestive heart failure
* No significant arrhythmias
* No myocardial infarction within the past 3 months
* No unstable angina pectoris
* No unstable or uncompensated cardiac disease
* No other significant heart disease

Pulmonary

* No unstable or uncompensated respiratory disease

Immunologic

* No known severe hypersensitivity to ketoconazole or calcitriol or any of the excipients of these products
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to the study drugs
* No ongoing or active infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 3 months after completion of study treatment
* Able to receive oral medication
* No sperm donation during and for ≥ 3 months after completion of study treatment
* No evidence of significant clinical disorder or laboratory finding that would preclude study participation
* No other severe or uncontrolled systemic disease
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic growth factors, including filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

  * Any number of prior chemotherapy regimens allowed

Endocrine therapy

* No concurrent systemic glucocorticoid therapy > physiologic replacement doses

Radiotherapy

* See Disease Characteristics
* Any number of prior radiotherapy regimens allowed

Surgery

* See Disease Characteristics
* Recovered from prior major surgery
* Concurrent surgery allowed provided ≥ 7 days has passed since the last dose of ketoconazole (ketoconazole may be restarted after adequate wound healing)

Other

* Recovered from prior anticancer therapy

  * Alopecia allowed
* More than 30 days since prior nonapproved or investigational agents
* More than 7 days since prior and no concurrent thiazides
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent digoxin or calcium supplementation
* No concurrent proton pump inhibitor or H2 blockers
* No concurrent medications that would alter the levels of ketoconazole and/or calcitriol, including the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates (e.g., phenobarbital)
  * Rifampin
  * Hypericum perforatum (St. John's wort)
* No concurrent drugs that would be significantly impaired in a clinically important way by ketoconazole
* No other concurrent investigational or commercial agents or therapies for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-11; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of calcitriol

SECONDARY OUTCOMES:
Pharmacokinetics of calcitriol and dexamethasone with or without ketoconazole

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States